CLINICAL TRIAL: NCT02388672
Title: Evaluation of Effects of Green Coffee Bean Extract (GCE) on Physiological and Psychological Variables- a Randomized, Placebo-controlled and Double-blinded Study in Healthy Subjects
Brief Title: Evaluation of Effects of Green Coffee Bean Extract (GCE) on Physiological and Psychological Variables
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel changes
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Isabelle Mack, Dr., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GCB1
Record Dates: First submitted 2015-02-19; First posted 2015-03-17 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Chlorogenic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Drink high-CGA (Experimental): Participants will drink once 250ml of decaffeinated coffee enriched with chlorogenic acid (CGA) (6g decaffeinated coffee (5 mg caffeine) with high total CGA (560 mg)).
  Interventions: Dietary Supplement: decaffeinated coffee; Dietary Supplement: chlorogenic acid
- Drink low-CGA (Placebo Comparator): 6g decaffeinated coffee (250 ml) with normal total CGA (224 mg)
  Interventions: Dietary Supplement: decaffeinated coffee; Dietary Supplement: chlorogenic acid
- Capsules high-CGA (Experimental): 6g decaffeinated coffee (250 ml) with normal total CGA and 800mg green coffee bean extract supplement with total CGA (560mg)
  Interventions: Dietary Supplement: decaffeinated coffee; Dietary Supplement: chlorogenic acid; Dietary Supplement: green coffee bean extract supplement
- Capsules low-CGA (Placebo Comparator): 6g decaffeinated coffee (250 ml) with normal total CGA and placebo
  Interventions: Dietary Supplement: decaffeinated coffee; Dietary Supplement: chlorogenic acid; Dietary Supplement: placebo
- Control (No Intervention): No treatment control group

INTERVENTIONS:
Dietary Supplement: decaffeinated coffee — Decaffeinated coffee with low chlorogenic acid (224mg; low-CGA)
  Arms: Capsules high-CGA; Capsules low-CGA; Drink high-CGA; Drink low-CGA
Dietary Supplement: chlorogenic acid — Decaffeinated coffee with high chlorogenic acid (560mg; high-CGA)
  Arms: Capsules high-CGA; Capsules low-CGA; Drink high-CGA; Drink low-CGA
Dietary Supplement: green coffee bean extract supplement — Decaffeinated coffee together with green coffee bean extract supplement (560mg; high-CGA)
  Arms: Capsules high-CGA
Dietary Supplement: placebo — Decaffeinated coffee with placebo capsules as control group for green coffee bean extract supplement (224mg; low-CGA)
  Arms: Capsules low-CGA

SUMMARY:
Coffee as one of the most favorite worldwide beverages comprises a variety of chemicals with health benefits. Most investigations have so far focused on the beneficial effects of caffeine but knowledge about non-caffeine coffee compounds such as chlorogenic acid (CGA) is scarce. The reducing risk of a variety of diseases following CGA consumption has been mentioned in recent basic and clinical studies. However, there is a lack of studies that examine the behavioral effects of CGA. This study aims to fill this gap.

In a randomized double-blind study, the investigators test the acute effects of coffee enriched with CGA or CGA supplement on physiological functions such as blood pressure, blood glucose, and heart rate, and on psychological functions such as mood and cognitive performance in 30 healthy adult subjects (18-40 years).

Participants will be allocated to an intervention plan using computer-generated random numbers. Treatments comprise of (1) 6g decaffeinated (5 mg caffeine) coffee (250 ml) with high total CGA (560 mg), or (2) 6g decaffeinated coffee (250 ml) with normal total CGA (224 mg), or (3) 6g decaffeinated coffee (250 ml) with normal total CGA and 800mg green coffee bean extract with total CGA (560mg), or (4) 6g decaffeinated coffee (250 ml) with normal total CGA and placebo, or (5) no treatment group. Upon arrival in the laboratory, participants will complete a 24-hour food recall, a psychometric test battery, and mood and cognitive performance tests. The tests will be repeated 40 min following CGA application, which coincide with the approximated peak of CGA blood concentrations and at 120 min post treatment. Blood pressure, blood glucose and heart rate recordings will be taken prior to treatment and at 1, 30, 60, 90 and 120 min post-treatment. The response to GCE-enriched coffee will be compared to GCE supplement for each of the groups of variables.

DETAILED DESCRIPTION:
Coffee as one of the most favorite worldwide beverages comprises a variety of chemicals maintaining the greatest health benefits among the commonly consumed beverages. Most investigations have so far focused on the beneficial effects of caffeine. On the contrary, knowledge on potential health benefits of non-caffeine coffee compounds is scarce. Coffee contains many polyphenols, especially chlorogenic acids (CGA), which have purported antioxidant abilities. With increasing incidence of degenerative diseases, the general public is turning to use natural herbal supplements, as one of these agents, CGA has been biologically and medically emphasized and can be expected to become a topic addressed in future studies, medical trends and pharmacology. The reducing risk of a variety of diseases following CGA consumption has been mentioned in recent basic and clinical studies. However, there is a lack of studies that examine the behavioral effects of CGA. This study aims to fill this gap.

In a randomized double-blind study, the investigators test the acute effects of coffee enriched with CGA or CGA supplement on physiological functions such as blood pressure, blood glucose, and heart rate, and on psychological functions such as mood and cognitive performance in 30 healthy adult subjects (18-40 years).

Participants will be allocated to an intervention plan using computer-generated random numbers. Treatments comprise of (1) 6g decaffeinated (5 mg caffeine) coffee (250 ml) with high total CGA (560 mg), or (2) 6g decaffeinated coffee (250 ml) with normal total CGA (224 mg) , or (3) 6g decaffeinated coffee (250 ml) with normal total CGA and 800mg green coffee bean extract with total CGA (560mg), or (4) 6g decaffeinated coffee (250 ml) with normal total CGA and placebo, or (5) no treatment group. Participants will be instructed to abstain from alcohol, foods, and beverages containing caffeine, chlorogenic acids and high polyphenol content for 24 hours prior to the experiment. Upon arrival in the laboratory, participants will complete a 24-hour food recall, a psychometric test battery consisting of the questionnaire on competence and control beliefs (FKK), the Life Orientation Test-Revised (LOT-R), the Beliefs about Medicines Questionnaire (BMQ), the Sensitivity to Punishment and Reward Questionnaire (SPSRQ), General Self-Efficacy (SWE) questionnaire, and mood and cognitive performance tests consisting of the Profile of Mood States (POMS) questionnaire, a parametric Go/no-Go test (PGNG) and the California Verbal Learning Test (CVLT). The POMS, Go/no-Go, and CVLT will be repeated 40 min following CGA application, which coincide with the approximated peak of CGA blood concentrations and at 120 min post treatment. Blood pressure, blood glucose and heart rate recordings will be taken prior to treatment and at 1, 30, 60, 90 and 120 min post-treatment. The response to GCE-enriched coffee will be compared to GCE supplement for each of the groups of variables.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 40 years old
* Normal weight (BMI > 18 and < 25 kg/m2)
* Regular coffee drinkers (1 to 2 cups/day)
* Both male and female

Exclusion Criteria:

* BMI <18 or >25 kg/m2
* Systolic blood pressure (SBP) <100 or >160 mmHg
* Diastolic blood pressure (DBP) <50 or >100 mmHg
* History of neurological, psychiatric, cardiac, endocrine or other disorders
* History of substance abuse
* Current use of antihypertensive and psychotropic medication
* More than 30 g/day alcohol consumption
* Woman who are pregnant or lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
blood pressure | from baseline to 30 min after intake of CGA

SECONDARY OUTCOMES:
heart rate | from baseline to 30 min after intake of CGA
blood glucose | from baseline to 30 min after intake of CGA
mood (Profile of Mood States (POMS) questionnaire) | from baseline to 30 min after intake of CGA
  Assessed with the Profile of Mood States (POMS) questionnaire
cognitive performance (parametric go/no-go task) | from baseline to 30 min after intake of CGA
  Assessed with a parametric go/no-go task measuring reaction times, attention (percentage of correct trials), and inhibition (percentage of correct inhibited trials)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mack, Dr., Principal Investigator — University Hospital Tübingen